CLINICAL TRIAL: NCT06862492
Title: Comparing Open Surgical, Modified Seldinger's and Ultrasound Guided Techniques for Jugular Central Line Insertion in Infants
Brief Title: Open Surgical, Modified Seldinger's and US Techniques for Jugular Central Line Insertion in Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Salah Eldin Amin, Demonstrator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264MS38/1/23
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Infants; Intensive Care Unit; Central Venous Catheterization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open surgical technique group (Experimental): included 35 patients underwent Central venous catheterization insertion using Open surgical technique group
  Interventions: Device: Open surgical cut down technique
- Modified Seldinger's technique group (Experimental): included 35 patients underwent Central venous catheterization insertion
  Interventions: Device: Modified Seldinger's technique
- Ultrasound guided Central venous catheterization insertion group (Experimental): included 35 patients underwent closed ultrasound guided Central venous catheterization insertion
  Interventions: Device: Closed Ultrasound guided CVC insertion

INTERVENTIONS:
Device: Open surgical cut down technique — The technique was performed following the descriptions of Farhadi et al. The infant was positioned in 30° (Trendelenburg's position), with a roll under his shoulders for neck extension and rotated to contralateral side of the surgical side to expose the incision site. Incision was done under sedation and pulse oximeter to monitor the oxygen saturation during the technique.
  Under complete aseptic technique, a small transverse incision 1cm was made on triangle bordered by the clavicle inferiorly and by the sternal and clavicular heads of the sternomastoid muscle medially and laterally. With blunt dissection we separate the two heads of the sternomastoid exposing the internal jugular vein .
  Then internal jugular vein cut down was performed and catheter inserted through it, all internal jugular vein venotomies were repaired as needed by 6/0 Polypropylene (Prolene®) suture and the wound was closed by absorbable polyglactin (Vicryl) suture
  Arms: Open surgical technique group
Device: Modified Seldinger's technique — After proximal and distal control of the vein, a 24-G. cannula was carefully inserted directly to the internal jugular vein . The guidewire was inserted through the cannula, then the cannula was removed. A size 4-5 French short length catheter was passed and brought out through the guidewire, then the guidewire was removed. The wound was closed after the correct catheter position and good haemostasis was obtained; the area was covered with sterile dressing.
  Arms: Modified Seldinger's technique group
Device: Closed Ultrasound guided CVC insertion — Ultrasound probe was connected to ultrasound unit and focused with ultrasonic gel and wrapped in a sterile plastic sheath. By wrapping the transducer in a sterile sheath, the probe place perpendicular to the long axis of the vessel, standard US two-dimensional (2D) imaging was used to visualize the vein in the short-axis view as a circle. Catheterization was performed under continuous dynamic observation of real-time 2D images. Insertion needle was advanced through the skin under US guidance into the internal jugular vein . A guidewire was then placed through the needle into the vein, and the needle was removed. Then catheter was inserted over the wire into internal jugular vein .
  Arms: Ultrasound guided Central venous catheterization insertion group

SUMMARY:
The aim of this study was to compare the three approaches: open technique, modified Seldinger's technique and closed ultrasound-guided Central venous catheterization insertion for central line insertion in infancy as regards safety, success of cannulation, technique time, and preservation of the patency of the internal jugular vein.

DETAILED DESCRIPTION:
Central venous catheterization is an essential technique in the intensive care units , for the administration of life-saving treatments including total parenteral nutrition, nutritional support, and intravenous medication. The internal jugular vein is often chosen because of its relatively larger size than the subclavian vein, lower risk of complications, and easy compressibility in case of bleeding. To facilitate Central venous catheterization, ultrasound guidance over anatomical guidance in closed techniques has been introduced bringing increased success rates, decreased catheterization times, and reduced complications.

Open surgical insertion is a common method of tunneled catheter implantation in the past, but the percutaneous approach has recently gained more popularity . The modified Seldinger's insertion technique is a catheter over guide wire technique, based on the original Seldinger's technique, and has not been widely adopted in Intensive care units. However, the modified Seldinger's technique has been successfully introduced into Intensive care units, and it is now used as the only technique for peripherally inserted central venous catheter insertion .

Central venous catheterization have become a mandatory part of clinical management in a variety of clinical circumstances in pediatric age groups. It allows resuscitation for intravascular fluid depletion and access for vasoactive medications and antibiotics, and it provides a means for hemodynamic monitoring and pacing. US guided closed technique is the updated use for insertion of IJV catheterization because it can both increase the success rate and decrease the complications related to Central venous catheterization placement

ELIGIBILITY:
Inclusion Criteria:

- 1-patients needed Central venous catheterization insertion in the internal jugular vein for medical or surgical causes.

2- patients with age ranging from birth till two years

Exclusion Criteria:

* 1- femoral or subclavian Central venous catheterization insertion. 2- patients with thrombosed internal jugular vein . 3- patients with previous Central venous catheterization insertion. 4- those with malignant conditions

Ages: 1 Hour to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2025-08-21 (Estimated); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-08-21 (Estimated)

PRIMARY OUTCOMES:
success of cannulation | 20 minutes
  Central venous cannulations in pediatric patients using each technique

SECONDARY OUTCOMES:
Technique time | within 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Amin, Demonstrator, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from principle investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For one year
Access Criteria: Statistical analysis was done using Statistical Package for the Social Sciences (SPSS) v27 (IBM©, Armonk, IL, USA). The Shapiro-Wilks test and histograms were used to evaluate the normality of the distribution of data. Quantitative parametric data were presented as mean and standard deviation (SD) and were analysed by one way ANOVA (F) test with post hoc test (Tukey). Quantitative non-parametric data were presented as median and interquartile range (IQR) and were analysed using Kruskal-Wallis test and/or Mann Whitney-test to compare each group. Qualitative variables were presented as frequency and percentage (%) and were analyzed utilizing the Chi-square test. A two tailed probability (P) value <0.05 was considered statistically significant.

REFERENCES:
- [Derived] Salah Eldin MM, Shehata SMK, Shehata MA, Elhaddad AA. Comparing open surgical, SELDINGER'S technique with surgical isolation of the vein and ultrasound guided techniques for jugular central line insertion in infants: a randomized clinical trial. BMC Surg. 2025 Jul 3;25(1):280. doi: 10.1186/s12893-025-02988-5. PMID 40611041